CLINICAL TRIAL: NCT07067580
Title: Effect of Breathing Exercise on Pain and Quality of Recovery in After Transplantation Patients: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Tuba Yılmazer, Principal investigator, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: transplantationsurgery
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Transplantation; Pain Management; Quality of Recovery 40
MeSH Terms: conditions — Agnosia | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): After obtaining permission from the experimental group with the "Informed Consent Form" the day before the surgery, the patients who agree to participate in the study will fill out the "Patient Introduction Form" by the researchers. The respiratory exercises will be taught and monitored by the researchers, and the researcher who will perform them works as a nurse in the general surgery department. The experimental group will be trained on respiratory exercises by the researcher the day before the surgery. The patients will be asked to perform the post-operative respiratory exercises as 1 set (4 breaths) per hour. The patient's vital signs will be monitored before and after the respiratory exercise. Patients will not have difficulty during the respiratory exercise, they will be asked to do it gradually. Pain conditions will be monitored at 0, 2, 6, 12 and 24 hours during the 24-hour hospital stay. The recovery quality scale will be applied on the 1st and 3rd days after the surgery.
  Interventions: Other: respiratory exercise
- Control (No Intervention): In the control group, after obtaining permission with the "Informed Consent Form" the day before the surgery, the patients who agreed to participate in the study will fill out the "Patient Introduction Form" by the researchers, and their pain status will be monitored at 0, 2, 6, 12 and 24 hours during the 24-hour hospital stay after the surgery. The quality of recovery scale will be applied on the 1st and 3rd days after the surgery. No intervention will be made to the patients in the control group, and they will receive routine nursing care provided in the hospital.

INTERVENTIONS:
Other: respiratory exercise — The experimental group will be trained on respiratory exercises by the researcher the day before the surgery. The patients will be asked to perform the post-operative respiratory exercises as 1 set (4 breaths) per hour. The patient's vital signs will be monitored before and after the respiratory exercise. Patients will not have difficulty during the respiratory exercise, they will be asked to do it gradually.
  Arms: Experimental

SUMMARY:
The researchers will fill out the "Patient Introduction Form" for the patients who agreed to participate in the study after obtaining permission from the experimental group with the "Informed Consent Form" the day before the surgery. The breathing exercises will be taught and monitored by the researchers, and the researcher who will implement them is a nurse in the general surgery department. The experimental group will be trained on breathing exercises by the researcher the day before the surgery. The patients will be provided with 1 set (4 breaths) per hour of breathing exercises after the surgery. The patient's vital signs will be monitored before and after the breathing exercise. Patients will not have difficulty during the breathing exercise, and they will be provided with gradual interventions. Pain status will be monitored at 0, 2, 6, 12 and 24 hours during the 24-hour hospital stay. The recovery quality scale will be applied on the 1st and 3rd day after surgery. In the control group, after obtaining permission with the "Informed Consent Form" the day before the surgery, the patients who agreed to participate in the study will fill out the "Patient Introduction Form" by the researchers, and their pain status will be monitored at 0, 2, 6, 12 and 24 hours during the 24-hour hospital stay after the surgery. The recovery quality scale will be applied on the 1st and 3rd day after surgery. No intervention will be made to the patients in the control group, and they will be provided with routine nursing care provided in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over, 65 and under,
* Those who have had a transplant for the first time,
* Patients who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Hemodynamically unstable,
* Those who may experience physical strain during breathing exercises and have a disease that may cause increased intra-abdominal pressure (e.g. bleeding hemorrhoids, hernias of all kinds, persistent cough, severe back pain, heart diseases, high blood pressure, urinary incontinence, epilepsy),
* Those with early complications
* Those with neurological or psychological problems,
* Those who were transferred to the intensive care unit after surgery,
* Emergency and unplanned cases will be excluded from the scope of the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
visual analog scale | postoperative 2,6,12,24 hours
  The scale consists of a 10 cm long horizontal line and the score is determined by measuring the distance between the leftmost end of the scale and the point marked by the patient. The score range from 0 to 10 on this scale and higher scores indicate increased pain severity.
Quality of Recovery-40 | postoperative 1 and 3 days
  It was developed by Myles et al. (2000) and its Turkish validity and reliability were conducted by Karaman et al. (2014). The questionnaire consists of 40 items and five sub-dimensions as 'Emotional State, Physical Comfort, Patient Support, Physical Independence, and Pain'. Each item in the questionnaire is scored on a Likert-type scale ranging from 1 to 5. This classification is as follows: 1= Never, 2= Sometimes, 3= Usually, 4= Most of the time, 5= Always. The total score obtained from the scale varies between 40 and 200. An increase in the score obtained from the questionnaire indicates that the physical and emotional well-being of the patients increases in the postoperative period; a decrease indicates that the physical and emotional well-being of the patients is negatively affected (Myles et al. 2000; Karaman et al. 2014). The Cronbach's alpha coefficient of the questionnaire was determined as 0.936 (Karaman et al. 2014).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)